CLINICAL TRIAL: NCT00470613
Title: A Phase I Open-Label Safety and Pharmacokinetic Study of Escalating Doses of SGT-53 for Infusion in Subjects With Advanced Solid Tumors
Brief Title: Safety Study of Infusion of SGT-53 to Treat Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SynerGene Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGT53-01
Record Dates: First submitted 2007-05-04; First posted 2007-05-08 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Neoplasm
Keywords: Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SGT-53 (Experimental): SGT-53 (2.4mg DNA/infusion) will be administered in a standard 3x3 dose escalation design in combination with docetaxel 40mg/m2 starting dose, cohort 1, cycle 1. This protocol will allow for both inter- and intra-patient dose escalations. SGT-53 will be administered weekly, day 1 except weeks 1, 4 & 7 when it will be administered biweekly on days 1 & 4. Docetaxel will be administered every 3 weeks (weeks 1, 4 & 7) on day 3. Patients completing cohort 1, cycle 1 without DLT at docetaxel 40mg/m2 will be allowed to dose escalate to 60mg/m2 in cycles 2 and 3. Cohort 2 (2.4mg DNA/infusion;75mg/m2 Docetaxel) will open 3 weeks after demonstration of 0/3 or ≤1/6 DLTs at docetaxel 60mg/m2. Cohort 3 (3.6mg DNA/infusion; 75mg/m2 Docetaxel) will open after demonstration of 0/3 or ≤1/6 DLTs at SGT-53 2.4mg DNA/infusion and docetaxel 75mg/m2. If necessary, the dose of docetaxel in cycle 2 and 3 may be reduced to 60mg/m2.
  Interventions: Genetic: SGT-53

INTERVENTIONS:
Genetic: SGT-53 — For Phase Ib: SGT-53 (2.4 mg DNA per infusion) will be administered in combination with docetaxel at 40 mg/m2 starting dose, cohort 1, cycle 1. SGT-53 will be administered weekly, on day 1 in weeks 2, 3, 5, and 6, and biweekly on days 1 and 4 in weeks 1, 4, and 7. Docetaxel will be administered every 3 weeks (weeks 1, 4, and 7)on day 3. Patients completing cohort 1, cycle 1 without DLT at 40 mg/m2 docetaxel will be allowed to dose escalate to 60 mg/m2 docetaxel in cycles 2 and 3.Cohort 2 (2.4mg DNA/infusion;75mg/m2 Docetaxel) will open 3 weeks after demonstration of 0/3 or ≤1/6 DLTs at docetaxel 60 mg/m2. Cohort 3 (3.6 mg DNA/infusion; 75 mg/m2 Docetaxel) will open after demonstration of 0/3 or ≤1/6 DLTs at SGT-53 2.4 mg DNA/infusion and docetaxel 75 mg/m2.

SUMMARY:
This is a Phase Ib study as a continuation of the original Phase I protocol. The purpose of this Phase Ib study is to evaluate the safety of a single course of SGT-53 in combination with docetaxel and determine the recommended Phase II doses of SGT-53 and docetaxel in combination for evaluation in subsequent clinical studies for the treatment of solid tumors.

DETAILED DESCRIPTION:
The p53 gene is a vital tumor suppressor gene in humans. Numerous human tumors possess a loss or mutation of wild type p53 (wtp53). In addition to playing a crucial role in cell cycle control, the p53 gene is a critical component in two of the pathways involved in regulating tumor cell growth: cell death (apoptosis) and the regulation of angiogenesis. The loss of such critical tumor suppressor activity is believed to be responsible for p53's involvement in such a broad array of human tumors and resistance to chemo/radiotherapy. SGT-53 is a complex composed of a wild type p53 gene (plasmid DNA) encapsulated in a liposome that is targeted to tumor cells by means of an anti-transferrin receptor single-chain antibody fragment (TfRscFv) attached to the outside of the liposome. Pre-clinical studies have indicated that SGT-53 could sensitize tumors to the effects of radiation/chemotherapy.

The Phase 1a portion of this clinical study was designed to evaluate the safety and maximum tolerated dose (MTD) of SGT-53. In addition, pharmacokinetics of escalating doses of SGT-53 will be measured and correlated with tumor response and toxicity.

The Phase Ib portion of this clinical study is designed to evaluate the safety of SGT-53 in combination with docetaxel, determine the recommended Phase II doses of these two agents, and evaluate the effect of the combination of SGT-53 and docetaxel on tumor size or progression.

ELIGIBILITY:
Inclusion Criteria:

* Have a biopsy confirmed diagnosis thereby providing histological diagnosis of a solid tumor malignancy.
* Have been offered all standard or approved therapies for which they would be considered eligible and have specifically declined or decided to postpone.
* Have solid tumors that can be measured on physical examination or by radiographic imaging studies.
* Have a tumor for which docetaxel would be an appropriate therapeutic agent (Phase Ib only).
* Patients (n=3) entered in phase Ib MTD dose expansion require biopsy accessible lesion in addition to measurable lesion and must consent to biopsy of tumor and normal skin.
* Previous docetaxel allowed if > 6 months prior to study entry (Phase Ib only).
* Be 18 years old or older.
* Have an ECOG performance study of 0, 1 or 2 for Phase Ia, 0-1 for Phase Ib.
* Be able to give informed consent.
* Have recovered from any previous therapy side effects or toxicities prior to initiating protocol study infusions.
* Have a life expectancy of more than 12 weeks.
* Female subjects of childbearing potential must have a negative pregnancy test within 7 days before initiation of study drug dosing. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Male and female subjects of reproductive potential must agree to use measures (e.g., condoms or birth control pills) to avoid pregnancy throughout the study and for 3 months following discontinuation of the study drug.
* Organ function characterized by </= Grade 1 scores defined by CTCAE v3.0 unless, at the discretion of the investigator, the condition is not deemed to cause unacceptable risk to the patient. If deemed not to cause unacceptable risk to the patient, organ function of grade 2 is acceptable.
* Laboratory values meeting the following criteria:

  * Hemoglobin >/= 10.0 gm/dL
  * Absolute neutrophil count > 1500/mm3
  * White blood cell count > 3000/mm3
  * Platelet count >/= 100,000/mm3
  * PT/PTT < 1.5 times the upper limit of normal
  * LDH </= 3 times the upper limit of normal and without clinical or laboratory evidence of DIC as determined by the clinical investigator
  * Total bilirubin </= 1.5 times the upper limit of normal (unless elevation is known to be due to Gilbert's Disease)
  * AST and ALT < 2.5 times the upper limit of normal withALP </= 2.5 x ULN
  * Creatinine </= 1.5 mg/dL or creatinine clearance >/= 50 ml/minute

Exclusion Criteria:

* Have hematological malignancy
* Prior hypersensitivity reaction to docetaxel (Phase Ib only)
* Are pregnant or lactating women
* Have signs and symptoms consistent with an active infection
* Fever (> 38.1 C)
* Treated with antibiotics for infection within one-week prior to study entry
* Known HIV infection
* Have any history of psychiatric disorders that would interfere with informed consent or follow-up.
* Have any other concurrent disease that, in the judgment of the investigator, would contraindicate the administration of study drug or interfere with the study evaluations.
* Have fasting glucose levels >/= 180 mg/dL.
* Have diastolic blood pressure of > 90 mm Hg resting at baseline despite medication. (Acceptable if on hypertensive medication and diastolic blood pressure is </= 90 mm Hg.)
* Have an abnormal stress echo or unfavorable results (at the discretion of the cardiologist) from the cardiac consultation and evaluation.
* Have known cardiac disease, or a history of cardiac disease.
* Had within six months prior to enrollment any of the following:

  * Cerebrovascular accident
  * Uncontrolled congestive heart failure (dyspnea on minimal exertion or while supine)
  * Unstable angina (chest pain greater than three times weekly while on therapy)
* Have significant baseline neuropathies (>/= grade 2 based upon CTCAE v 3.0).
* Requiring renal dialysis.
* Receiving systemic steroids or other chronic immunosuppressive medications (e.g., tacrolimus, cyclosporine) within 30 days prior to study entry
* Receiving hematopoietic growth factors
* Receiving anticoagulants other than to maintain patency of venous access lines
* Received an investigational drug within 30 days prior to study entry
* Received radiation treatment < 4 weeks prior to study entry
* Had prior exposure to gene vector delivery products within the last 6 months
* Received treatment with chemotherapeutic agents < 4 weeks prior to study entry except for mitomycin C or nitrosurea where subjects who received mitomycin C or nitrosoureas < 6 weeks prior to study entry are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Safety will be assessed by analysis of adverse experiences, clinical laboratory tests, and physical examinations. | 7 weeks

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 6 weeks
  Phase Ia Only
Tumor Response | Week 6 for Phase Ia, and weeks 9 for Phase Ib
  Assessed by physical measurements or by radiographic modalities
Determine the presence of exogenous wtp53 in tumor | Week 5 or Week 6

CONTACTS AND LOCATIONS:
Overall Officials: John J. Nemunaitis, MD, Principal Investigator — Mary Crowley Medical Research Center
Locations (1):
- Mary Crowley Medical Research Center, Dallas, Texas, United States